CLINICAL TRIAL: NCT02457221
Title: A Phase III, Randomized, Open, Parallel-controlled, Multi-center Study to Compare the Efficacy and Safety of Tacrolimus Capsules and Cyclophosphamide Injection in Treatment of Lupus Nephritis
Brief Title: A Study to Compare the Efficacy and Safety of Tacrolimus Capsules and Cyclophosphamide Injection in Treatment of Lupus Nephritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F506-CL-0912
Record Dates: First submitted 2015-05-22; First posted 2015-05-29 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Lupus Nephritis
Keywords: Tacrolimus; Cyclophosphamide; Prograf; lupus nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Tacrolimus; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tacrolimus group (Experimental): Tacrolimus capsules + steroid
  Interventions: Drug: Tacrolimus capsules; Drug: Prednisone
- Cyclophosphamide group (Active Comparator): Cyclophosphamide injections + steroid
  Interventions: Drug: Cyclophosphamide injections; Drug: Prednisone

INTERVENTIONS:
Drug: Tacrolimus capsules — oral
  Other Names: Prograf
  Arms: Tacrolimus group
Drug: Cyclophosphamide injections — intravenous injection
  Arms: Cyclophosphamide group
Drug: Prednisone — oral

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of Tacrolimus capsules for induction remission in patients with lupus nephritis, and compare the efficacy and safety with Cyclophosphamide injections.

DETAILED DESCRIPTION:
This is a randomized, open, 1:1 parallel controlled, multi-center, non-inferiority clinical study.

ELIGIBILITY:
Inclusion Criteria:

* 18.5≤Body Mass Index (BMI) <27;
* Diagnosed as systemic lupus erythematosus (based on American Rheumatism Association Diagnostic Criteria 1997)
* Diagnosed as III, IV, V, III + V, IV + V lupus nephritis (according to the LN classification in International Society of Nephrology and Renal Pathology Society (ISN/RPS) 2003) within 24 weeks before enrollment with renal biopsy;
* 24-hour urine protein ≥ 1.5g, Scr<260umol/L (or 3mg/dL)

Exclusion Criteria:

* Class II or VI lupus nephritis or renal biopsy chronic index (CI) > 3 or with TMA;
* Received immunosuppressants (mycophenolate mofetil (MMF), cyclosporine, methotrexate, mechlorethamine, chlorambucil, tripterygium preparations, leflunomide etc.) treatment with a duration of more than one week within 30 days prior to enrollment;
* Received tacrolimus (except for topical use) or cyclophosphamide treatment within 30 days prior to enrollment;
* Received a course of methylprednisolone (MP) pulse therapy or gamma globulin treatment or plasma exchange within 30 days prior to enrollment;
* Patients with history of allergies to tacrolimus, cyclophosphamide or methylprednisolone;
* Pregnancy, lactation or patient unwilling to take contraceptive measures;
* Patients with estimated maintenance dialysis for more than eight weeks; or dialysis for more than two weeks prior to entering observation;
* Patients received kidney transplantation or plan to have kidney transplantation recently;
* Serum creatinine (Scr) ≥260umol/L (or 3mg/dL) or creatinine clearance rate (Ccr) < 30ml/(min.1.73m2); according to Cockcroft-Gault formula: Ccr (ml/sec) = [(140- age)× Weight (kg)] × K / [72×Scr (umol/L) ×0.6786], Female K = 0.85, Male K = 1.0;
* Patients suffering from liver dysfunction (aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 3 times the upper limit of normal lab value) or bilirubin more than 3 times the upper limit of normal lab value;
* Patients diagnosed with diabetes;
* History of gastrointestinal bleeding or pancreatitis within 3 months;
* Uncontrollable hyperkalemia after dietary therapy or reduction of potassium treatment (exceed the upper limit of normal lab value);
* Patients suffering from lupus pneumonia or lung injury;
* Patients with anemia (hemoglobin <7g/dl) or bone marrow suppression (WBC <3.0×109/L, and/or neutrophils <1.5×109/L, and/or platelets <50×109/L) not secondary to systemic lupus erythematosus;
* With congenital heart disease, arrhythmia, heart failure or other severe cardiovascular diseases;
* With refractory hypertension (defined as blood pressure still exceeds 180/110 mmHg despite taking three different types of antihypertensive drugs [one of them is diuretic] simultaneously);
* Patients with recurrent tumors within 5 years;
* Severe infection that requires intravenous antibiotics within 2 weeks prior to enrollment;
* Patients with infection of hepatitis B virus or hepatitis C virus; patients with active tuberculosis; patients with severe immunodeficiency diseases (including active cytomegalovirus infection (positive CMV IgM antibody), or human immunodeficiency virus (HIV) infection, etc.);
* Patients with lupus encephalopathy or other life-threatening complication of systemic lupus erythematosus;
* Patients participated in other clinical trials within three months before enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 314 (Actual)
Dates: Start 2015-03-10 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Remission rate (complete remission + partial remission) | at 24 weeks
  complete remission: urine protein < 0.5g/24hr, and serum albumin≥3.5g/dl, and stable renal function (Scr increase ≤ 15% baseline value) partial remission: urine protein 0.5-3.5g/24hr (≥ 0.5 g/24hr and < 3.5 g/24hr), and urine protein decreased by >50% comparing with the baseline, and serum albumin ≥ 3.0g/dl, and stable renal function (Scr increase ≤ 15% baseline value)

SECONDARY OUTCOMES:
24-hour urine protein | at Day 1, Weeks 1, 2, 4, 8, 12, 16, 20, 24
Change of 24-hour urine protein from baseline | at Day 1, Weeks 1, 2, 4, 8, 12, 16, 20, 24
Serum albumin | at Day 1, Weeks 1, 2, 4, 8, 12, 16, 20, 24
Change of Serum albumin from baseline | at Day 1, Weeks 1, 2, 4, 8, 12, 16, 20, 24
Serum creatinine | at Day 1, Weeks 1, 2, 4, 8, 12, 16, 20, 24
Change of Serum creatinine from baseline | at Day 1, Weeks 1, 2, 4, 8, 12, 16, 20, 24
eGFR comparing with baseline | at Day 1, Weeks 1, 2, 4, 8, 12, 16, 20, 24
  eGFR: Estimated Glomerular Filtration Rate
Percentage of patients converted to other immunosuppressive therapy | during 24 weeks
Percentage of patients with serum creatinine rising to two times of the baseline | during 24 weeks
Percentage of patients with dsDNA and ANA converting from positive to negative | during 24 weeks
  ANA: Antinuclear Antibody
SLE-DAI | at Week 4, 12 and 24
  SLE-DAI: Systemic Lupus Erythematosus - Disease Activity Index
Immune parameters assessed by ESR, C3, C4 and dsDNA | at Week 4, 12 and 24
  ESR: Erythrocyte Sedimentation Rate, C3, C4: Complement C3, C4, dsDNA: Anti-Double-Stranded DNA Antibodies
Change of SLE-DAI from baseline | at Week 4, 12 and 24
Change of immune parameters from baseline | at Week 4, 12 and 24
Renal biopsy AI (Active Index) | at Week 24
CI (Chronic Index) | at Week 24
Change of Renal biopsy AI (Active Index) from baseline | at Week 24
Change of CI (Chronic Index) from baseline | at Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma China, Inc.
Locations (35):
- China (35):
  - Site CN00043, Hefei, Anhui
  - Site CN00030, Beijing, Beijing Municipality
  - Site CN00034, Beijing, Beijing Municipality
  - Site CN00041, Xiamen, Fujian
  - Site CN00056, Guangzhou, Guangdong
  - Site CN00017, Shenzhen, Guangdong
  - Site CN00045, Liuchow, Guangxi
  - Site CN00037, Nanning, Guangxi
  - Site CN00038, Nanning, Guangxi
  - Site CN00020, Shijiazhuang, Hebei
  - Site CN00047, Shijiazhuang, Hebei
  - Site CN00028, Zhengzhou, Henan
  - Site CN00023, Wuhan, Hubei
  - Site CN00024, Wuhan, Hubei
  - Site CN00027, Changsha, Hunan
  - Site CN00050, Changsha, Hunan
  - Site CN00012, Nanjing, Jiangsu
  - Site CN00013, Nanjing, Jiangsu
  - Site CN00025, Nanjing, Jiangsu
  - Site CN00049, Wuxi, Jiangsu
  - Site CN00026, Changchun, Jilin
  - Site CN00042, Changchun, Jilin
  - Site CN00005, Dalian, Liaoning
  - Site CN00018, Shenyang, Liaoning
  - Site CN00019, Shenyang, Liaoning
  - Site CN00032, Qingdao, Shandong
  - Site CN00001, Shanghai, Shanghai Municipality
  - Site CN00014, Shanghai, Shanghai Municipality
  - Site CN00015, Shanghai, Shanghai Municipality
  - Site CN00052, Taiyuan, Shanxi
  - Site CN00002, Chengdu, Sichuan
  - Site CN00003, Chengdu, Sichuan
  - Site CN00021, Tianjin, Tianjin Municipality
  - Site CN00044, Ürümqi, Xinjiang
  - Site CN00010, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Zheng Z, Zhang H, Peng X, Zhang C, Xing C, Xu G, Fu P, Ni Z, Chen J, Xu Z, Zhao MH, Li S, Huang X, Miao L, Chen X, Liu B, He Y, Li J, Liu L, Kadeerbai H, Liu Z, Liu Z. Effect of Tacrolimus vs Intravenous Cyclophosphamide on Complete or Partial Response in Patients With Lupus Nephritis: A Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e224492. doi: 10.1001/jamanetworkopen.2022.4492. PMID 35353167
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=381